CLINICAL TRIAL: NCT03993704
Title: A Double-blind, Placebo-controlled, Dose-escalation Study of the Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of LHF-535 (LHF-535-SDD) in Healthy Participants
Brief Title: Multiple Ascending Oral Dose 14-Day Trial of LHF-535 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kineta Inc. (Industry)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KVHF-535-102
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Lassa fever; viral hemorrhagic fever
MeSH Terms: conditions — Lassa Fever; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): 450 mg, 1125 mg, or 2250 mg of LHF-535 given once daily for 14 days
  Interventions: Drug: LHF-535
- Placebo (Placebo Comparator): Placebo to match LHF-535 given once daily for 14 days
  Interventions: Drug: LHF-535

INTERVENTIONS:
Drug: LHF-535 — Oral suspension administered once daily for 14 days

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of a daily oral dose of LHF-535 administered for 14 days to healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, multiple dose study to assess the safety, tolerability, and pharmacokinetics (PK) of multiple doses of orally administered LHF-535 in 24 to 32 healthy adult participants. Three successive escalating cohorts, each containing 8 participants, are planned. Within each cohort, 6 participants will be randomized to receive an oral dose of LHF-535 once daily for 14 days, and 2 will be randomized to receive an oral dose of placebo once daily for 14 days. After a screening period of up to 28 days, all participants will be confined to the study center from 1 day prior to dosing until at least 24 hours after the 14th day of dosing. Participants will return for follow-up evaluations on Day 17 and Day 21 (72 and 168 hours after last dose, respectively) and on Day 42. After each cohort, safety data through Day 17 and PK data through Day 7 will be reviewed by a blinded Safety Committee prior to dosing of the next cohort. The Safety Committee is charged with making one of the following three recommendations: (1) proceed with dose escalation as planned, (2) continue the study with modification (e.g., proceed with the next cohort at a lower dose level than planned), or (3) suspend the study. An additional cohort of 8 participants may be added to evaluate dosing for future studies, at the discretion of the Sponsor, in consultation with the Safety Committee.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 50 years of age, inclusive, at the time of screening
* Able to understand the requirements of the study, to provide written informed consent (as evidenced by signature on an informed consent document that is approved by a Human Research Ethics Committee [HREC]), and agreeable to abide by the study restrictions
* Body mass index (BMI) of 18.0 to 35.0 kg/m^2, inclusive, at the time of screening
* Weight between 50 kg and 110 kg, inclusive, at the time of screening and check-in (Day -1)
* Good general health (e.g., no chronic health conditions such as hypertension, diabetes, chronic obstructive pulmonary disease, or cardiovascular disease) as determined by the Investigator; participants with mild allergies or benign conditions such as Gilbert's disease may be enrolled at the discretion of the Investigator
* Female participants of child-bearing potential, with a fertile male sexual partner, must use a highly effective method of contraception (oral contraceptive, intrauterine device, or hormonal patch, injectable, or implantable device) in conjunction with a male condom during the screening period and for the entire duration of study participation including the 28-day follow-up; true abstinence from sexual intercourse with a partner of the opposite sex, in accordance with the preferred and usual lifestyle of the participant, is acceptable; periodic abstinence or avoiding sexual intercourse on days while the participant is fertile (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), are not acceptable methods of contraception; non-childbearing potential is defined as postmenopausal as documented by an elevated follicle stimulating hormone (FSH) level or surgical sterility (e.g., tubal ligation, hysterectomy, and/or bilateral salpingo-oophorectomy)
* Male participants must either be surgically sterile (vasectomy) or agree to use a male condom as a method of contraception for the entire duration of the study and for 90 days after dosing; the female sexual partner must also use a medically acceptable form of birth control (e.g., oral contraceptive)
* Male participants must agree to not donate sperm for the entire duration of the study and for at least 90 days after dosing

Exclusion Criteria:

* Pregnancy or breastfeeding
* A positive screen for drugs of abuse, including alcohol; the screen may be repeated once (on Day-1) at the Investigator's discretion if a false-positive result is suspected
* Use of more than 5 tobacco- or nicotine-containing products per week (including but not limited to: cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 3 months prior to check-in (Day -1) or use of tobacco- or nicotine-containing products within 72 hours of check-in (Day -1) until discharge from the study unit
* Donated blood within 90 days or plasma within 30 days of dosing on Day 1
* Any history of anaphylaxis to medication, food, animal toxin or other substances
* Active substance abuse or any medical or psychiatric condition that could jeopardize the participant's safety
* Use of any medications apart from vitamins, acetaminophen, or hormonal contraception within 14 days of dosing on Day 1 (unless approved by the Investigator and Sponsor Medical Monitor); participants with mild allergies may use antihistamines at the discretion of the Investigator after approval by the Sponsor Medical Monitor
* Receipt of an investigational product within 12 weeks prior to dosing on Day 1 (or 5 half-lives, whichever is longer)
* Any history of cancer; non-melanoma skin cancer or cervical cancer in situ, resected surgically with no evidence of disease, may be enrolled at the discretion of the Investigator
* Receipt of an organ transplant (solid or hematopoietic), including corneal transplant
* Prolonged QTcF interval >450 ms on electrocardiograms (ECGs) collected during screening, on Day -1, or just prior to dosing on Day 1 (following one repeat)
* Other clinically significant ECG abnormality, as determined by the Investigator
* Any clinically significant abnormal hematology, chemistry, or urinalysis value, as determined by the Investigator. Repeat testing is permitted at the discretion of the Investigator
* Positive test for human immunodeficiency virus (HIV serology) or known HIV infection
* Positive result for hepatitis B surface antigen (HBsAg) or for hepatitis C virus (HCV) antibody
* Use of alcohol-containing foods or beverages within 72 hours prior to check-in on Day -1 or 72 hours prior to any study visit
* Use of caffeine-containing foods or beverages within 24 hours prior to check-in on Day -1 until discharge from the study unit
* Strenuous exercise for 24 hours prior to check-in on Day -1 until discharge from the study unit
* Febrile illness or significant infection within 48 hours before administration of the first dose of study drug on Day 1

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events as Assessed by CTCAE v4.0 | 42 days
  Safety and tolerability

SECONDARY OUTCOMES:
Area Under the Plasma Concentration versus Time Curve (AUC) of LHF-535 | 21 days
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Studies, Melbourne, Australia